CLINICAL TRIAL: NCT00733291
Title: Evaluation of Daily Disposable Lenses With Multi-Purpose Solution (MPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MS-008
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Myopia
Keywords: Daily disposable contact lenses; Multi-purpose disinfecting solutions
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nelfilcon A soak / Nelfilcon A no-soak (Active Comparator): Nelfilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution, followed by nelfilcon A contact lenses inserted directly from the blister package. Each pair of lenses worn for 2 hours.
  Interventions: Device: Nelfilcon A contact lens; Device: FID 107027 solution
- Nelfilcon A no soak / nelfilcon A soak (Active Comparator): Nelfilcon A contact lenses inserted directly from the blister package, followed by nelfilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution. Each pair of lenses worn for 2 hours.
  Interventions: Device: Nelfilcon A contact lens; Device: FID 107027 solution
- Etafilcon A soak / etafilcon A no soak (Active Comparator): Etafilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution, followed by etafilcon A contact lenses inserted directly from the blister package. Each pair of lenses worn for 2 hours.
  Interventions: Device: Etafilcon A contact lens; Device: FID 107027 solution
- Etafilcon A no soak / etafilcon A soak (Active Comparator): Etafilcon A contact lenses inserted directly from the blister package, followed by etafilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution. Each pair of lenses worn for 2 hours.
  Interventions: Device: Etafilcon A contact lens; Device: FID 107027 solution

INTERVENTIONS:
Device: Nelfilcon A contact lens — Commercially marketed, single vision, soft contact lens for daily disposable wear
  Other Names: Focus Dailies with AquaRelease
  Arms: Nelfilcon A no soak / nelfilcon A soak; Nelfilcon A soak / Nelfilcon A no-soak
Device: Etafilcon A contact lens — Commercially marketed, single vision, soft contact lens for daily disposable wear
  Other Names: 1-Day ACUVUE Moist
  Arms: Etafilcon A no soak / etafilcon A soak; Etafilcon A soak / etafilcon A no soak
Device: FID 107027 solution — Commercially marketed solution for contact lens disinfection
  Other Names: Opti-Free RepleniSH Multi-Purpose Disinfecting Solution

SUMMARY:
The purpose of this study is to evaluate daily disposable lenses inserted out of the blister package versus daily disposable lenses inserted after a pre-soak in Multi-purpose solution FID 107027.

DETAILED DESCRIPTION:
Corneal staining and subjective responses for ocular redness and comfort will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Visual acuity correctable to 20/30 (Snellen) or better in each eye at distance with contact lenses.
* Successfully wearing hydrogel or silicone hydrogel contact lenses on a daily wear basis for at least two weeks prior to study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History of hypersensitivity to any components of the multi-purpose solution.
* Evidence or history of ocular conditions as prescribed in protocol.
* One functional eye or a monofit lens
* Any slit-lamp finding score equal to 1 at Visit 1 of each study period.
* Significant corneal staining at visit 1 of each study period as prescribed in protocol.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 subjects currently wearing hydrogel or silicone hydrogel lenses on a daily wear schedule for at least two weeks were enrolled between 1/7/08 and 2/1/08 by 4 US optometry sites
Pre-assignment Details: 18 hours of no contact lens wear (glasses only) served as the wash out before Period 1. This reporting group includes all enrolled and dispensed participants as treated.
Groups:
- Nelfilcon A Soak / Nelfilcon A no Soak; Etafilcon A Soak / Etafilcon A no Soak: Nelfilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution, followed by nelfilcon A contact lenses inserted directly from the blister package. Each pair of lenses worn for 2 hours.
- Nelfilcon A no Soak / Nelfilcon A Soak: Nelfilcon A contact lenses inserted directly out of the blister package, followed by nelfilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution. Each pair of lenses worn for 2 hours.
- Etafilcon A no Soak / Etafilcon Soak: Etafilcon A contact lenses inserted directly out of the blister package, followed by etafilcon A contact lenses inserted after being soaked overnight in a multi-purpose disinfecting solution. Each pair of lenses worn for 2 hours.
Period: First Intervention, 2 Hrs (+/- 30 Min)
Arm/Group | Nelfilcon A Soak / Nelfilcon A no Soak | Nelfilcon A no Soak / Nelfilcon A Soak | Etafilcon A Soak / Etafilcon A no Soak | Etafilcon A no Soak / Etafilcon Soak
Started | 13 | 17 | 17 | 17
Completed | 13 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period, 3 Days (+/-1 Day)
Arm/Group | Nelfilcon A Soak / Nelfilcon A no Soak | Nelfilcon A no Soak / Nelfilcon A Soak | Etafilcon A Soak / Etafilcon A no Soak | Etafilcon A no Soak / Etafilcon Soak
Started | 13 | 17 | 17 | 17
Completed | 12 | 17 | 17 | 17
Not Completed | 1 | 0 | 0 | 0
Not completed — Failed inc criteria Second Intervention | 1 | 0 | 0 | 0
Period: Second Intervention, 2 Hrs (+/- 30 Min)
Arm/Group | Nelfilcon A Soak / Nelfilcon A no Soak | Nelfilcon A no Soak / Nelfilcon A Soak | Etafilcon A Soak / Etafilcon A no Soak | Etafilcon A no Soak / Etafilcon Soak
Started | 12 | 17 | 17 | 17
Completed | 12 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A Contact Lens | Etafilcon A Contact Lens | Total
Number analyzed (Participants) | 29 | 34 | 63
Age, Categorical [Count of Participants; unit: Participants] — This reporting group is based on the number of subjects in the evaluable population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 27 | 34 | 61
    >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] — This reporting group is based on the number of subjects in the evaluable population.
  years | 37.59 (13.90) | 38.56 (12.42) | 38.11 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants] — This reporting group is based on the number of subjects in the evaluable population.
  Participants
    Female | 16 | 25 | 41
    Male | 13 | 9 | 22

OUTCOME MEASURES:

1. Secondary Outcome: Ocular Comfort
Description: Ocular comfort was recorded by the participant on a questionnaire using a 5-point scale. Participant completed the sentence, "Right now my eyes feel..." with one of the following responses: 1-very comfortable; 2-comfortable; 3-neither comfortable nor uncomfortable; 4-uncomfortable; 5-very uncomfortable.
Time Frame: After 2 hours of wear
Population: This reporting group is based on the number of subjects in the evaluable population for the indicated lens as treated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Nelfilcon A / FID 107027: Nelfilcon A contact lenses soaked overnight in multi-purpose disinfection solution (MPDS) prior to insertion
- Nelfilcon A / no Soak: Nelfilcon A contact lenses inserted directly out of the blister package
- Etafilcon A / FID 107027: Etafilcon A contact lenses soaked overnight in multi-purpose disinfection solution (MPDS) prior to insertion
- Etafilcon A / no Soak: Etafilcon A contact lenses inserted directly out of the blister package
Arm/Group | Nelfilcon A / FID 107027 | Nelfilcon A / no Soak | Etafilcon A / FID 107027 | Etafilcon A / no Soak
Number analyzed (Participants) | 29 | 29 | 34 | 34
Units on a scale | 1.86 (0.92) | 1.83 (0.80) | 1.65 (0.69) | 1.88 (0.88)

2. Primary Outcome: Average Corneal Staining Area
Description: Percentage corneal staining was assessed by the investigator for each of five regions of the cornea, i.e., four quadrants plus central. The investigator instilled fluorescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and a yellow filter. Percentage corneal staining area was recorded in increments of ten, and the percentages of the five regions were averaged together.
Time Frame: After 2 hours of wear
Population: This reporting group is based on the number of subjects in the evaluable population for the indicated lens as treated.
Measure: Mean (Standard Deviation); unit: Percentage area of cornea
Arm/Group | Nelfilcon A / FID 107027 | Nelfilcon A / No Soak | Etafilcon A / FID 107027 | Etafilcon A / no Soak
Number analyzed (Participants) | 29 | 29 | 34 | 34
Percentage area of cornea | 0.27 (0.39) | 0.08 (0.13) | 0.34 (0.63) | 0.18 (0.25)

3. Secondary Outcome: Ocular Redness
Description: Ocular redness was recorded by the participant on a questionnaire using a 5-point scale. Participant completed the sentence, "Right now my eyes look..." with one of the following responses: 1-very white; 2-white; 3-neither white nor red; 4-red; 5-very red.
Time Frame: After two hours of wear
Population: This reporting group is based on the number of subjects in the evaluable population for the indicated lens as treated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A / FID 107027 | Nelfilcon A / no Soak | Etafilcon A / FID 107027 | Etafilcon A / no Soak
Number analyzed (Participants) | 29 | 29 | 34 | 34
Units on a scale | 2.07 (0.46) | 2.10 (0.72) | 2.18 (0.76) | 2.06 (0.69)

4. Primary Outcome: Total Corneal Staining Type
Description: Total corneal staining type was assessed by the investigator for each of 5 regions of the cornea, i.e., four quadrants plus central. The investigator instilled fluorescein dye and examined the cornea with a slit lamp, i.e., biomicroscope and a yellow filter. Corneal staining type was recorded on a 5-point scale for each region: 0-none; 1-micropunctate; 2-macropunctate; 3-coalesced macropunctate; 4-patch (>/= 1mm). The five regions were summed.
Time Frame: After 2 hours of wear
Population: This reporting group is based on the number of subjects in the evaluable population for the indicated lens as treated.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A / FID 107027 | Nelfilcon A / no Soak | Etafilcon A / FID 107027 | Etafilcon A / no Soak
Number analyzed (Participants) | 29 | 29 | 34 | 34
Units on a scale | 1.59 (1.43) | 0.79 (1.18) | 1.32 (1.80) | 1.00 (1.23)

ADVERSE EVENTS:
Time Frame: For the duration of the study: 26 days.
Description: The safety population is defined as subjects who fulfilled the study entry criteria and had at least one insertion of a daily disposable study lens.
Groups:
- Etafilcon / no Soak: Etafilcon A contact lenses inserted directly out of the blister package
Arm/Group | Nelfilcon A / FID 107027 | Nelfilcon A / no Soak | Etafilcon A / FID 107027 | Etafilcon / no Soak
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party other than Contractors, the data arising out of the study.